CLINICAL TRIAL: NCT02949336
Title: Kinematics Analysis: Traditional (ACL Retaining) and ACL Deficient (Reduced Tibial Slope) Medial, Fixed Bearing Primary Unicondylar Knee Arthroplasty With the SIGMA® High Performance Partial Knee System
Brief Title: Kinematics Analysis of SIGMA® Partial Knee System
Acronym: UKA
Status: Completed | Type: Observational
Sponsor: Stephen Ferguson (Other)
Collaborators: Schulthess Klinik (Other); DePuy Synthes (Industry); Gelenkzentrum Zurich (Unknown)
Responsible Party: Sponsor-Investigator, Stephen Ferguson, Prof. Dr., Institute for Biomechanics, ETH Zürich
Organization: Institute for Biomechanics, ETH Zürich (Other)
Other Study IDs: UKA V 2.4 02.09.2016
Record Dates: First submitted 2016-10-24; First posted 2016-10-31 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Unicompartmental Knee Arthroplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Traditional UKA: Patients with a traditional Medial Unicompartmental Knee Arthroplasty, SIGMA® High Performance Partial Knee System (functional ACL and tibial posterior slope matching the native bone) will undergo observational use of fluoroscopy to analyze joint kinematics
  Interventions: Radiation: Observational use of fluoroscopy
- Group 2: ACL deficient UKA: Patients with the same medial UKA implant (SIGMA® High Performance Partial Knee System) in an ACL deficient knee, where the UKA was implanted at a 50% reduced tibial posterior slope relative to the native knee will undergo observational use of fluoroscopy to analyze joint kinematics.
  Interventions: Radiation: Observational use of fluoroscopy

INTERVENTIONS:
Radiation: Observational use of fluoroscopy — Minimal radiation exposure (0.17 mSv) for observational purpose

SUMMARY:
The proposed study is a prospective collection of health related personal data (observational study). A total of approximately 10 subjects with traditional medial SIGMA® High Performance Partial Knee System and 10 ACL deficient subjects with medial SIGMA® High Performance Partial Knee System are analyzed during sitting onto a chair and getting up, deep knee bend, stance and swing phase of level walking, downhill walking (ramp descent) and stair descent at least 12 months post-operatively, in terms of 3D fluoroscopic assessed tibio-femoral motion as well as simultaneous skin marker assessed whole leg motion and ground reaction forces. All the video-fluoroscopic testing is performed at the Institute for Biomechanics at the ETH Zurich. The UKA subjects are recruited based on the inclusion and exclusion criteria.

The primary objective is to quantify and describe the three-dimensional kinematics for patients with a traditional medial SIGMA® High Performance Partial Knee System (functional ACL and tibial posterior slope matching the native bone) during these daily activities.

The secondary objective is to evaluate patients with the same medial UKA implant (SIGMA® High Performance Partial Knee System) in an ACL deficient knee, where the UKA was implanted at a 50% reduced tibial posterior slope relative to the native knee.

DETAILED DESCRIPTION:
The knee arthroplasty for each patient was implanted more than one year ago as per inclusion criteria of this study with the sole purpose of standard clinical practice of the recruiting surgeons.

ELIGIBILITY:
Inclusion criteria (group 1):

* medial SIGMA® High Performance Partial Knee System due to medial OA
* Intact/functional ACL
* BMI ≤ 32
* good clinical outcome, KOOS >70
* no or very low pain VAS < 2
* Follow-up at least one year post-op
* Standardized general health survey score (SF-12) within the normal range for people in their age group
* Age ≥ 18 years

Exclusion criteria (group 1):

* Actual significant problem on lower extremities
* Misaligned UKA
* Deficient / non-functional ACL (Lachman Test)
* Any other arthroplasty at the lower extremities
* Patient incapable to understand and sign informed consent
* Incapable of performing the motion tasks
* Pregnancy

Inclusion criteria (group 2):

* medial SIGMA® High Performance Partial Knee System due to medial OA
* Deficient / non-functional ACL
* Central to posterior wear of medial tibial plateau (pre-op MRI)
* 50% reduced tibial posterior slope after UKA (post-op radiograph)
* BMI ≤ 32
* good clinical outcome, KOOS >70
* no or very low pain VAS < 2
* Follow-up at least one year post-op
* Standardized general health survey score (SF-12) within the normal range for people in their age group
* Age ≥ 18 years

Exclusion criteria (group 2):

* Actual significant problem on lower extremities
* Misaligned UKA / non-reduced posterior tibial slope (post-op radiograph)
* Intact / functional ACL
* Any other arthroplasty at the lower extremities
* Patient incapable to understand and sign informed consent
* Incapable of performing the motion tasks
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The clinical investigators of the participating clinics (PD Dr. med. Fabian von Knoch, Gelenkzentrum Zürich; and Dr. med. Stefan Preiss, Schulthess Klinik) will identify potential subjects based on clinical records. PD Dr. med. Fabian von Knoch will recruit patients he operated on at the Gelenkzentrum Zürich while Dr. med. Stefan Preiss will recruit subjects from his patient population at the Schulthess Klinik.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Knee Kinematics | 3 hours
  The primary outcome of this study is the relationship between the knee flexion angle and the medial and lateral anterior-posterior translation of the condyles during sitting onto a chair and getting up, deep knee bend, stance and swing phase of level walking, downhill walking (ramp descent) and stair descent.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ferguson, Prof. Dr., Study Director — Institute for Biomechanics, ETH Zurich
Locations (1):
- Institute for Biomechanics, ETH Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided